CLINICAL TRIAL: NCT00828945
Title: A Non-Randomized, Non-Controlled, Open Study In Order To Document The Compliance With Treatment, According To Clinical Praxis And National Guidelines For Patients With Hyperlipidemia. COLL: Control Of Lipid Lowering
Brief Title: Compliance With Treatment For Patients With Hyperlipidemia
Acronym: COLL
Status: Completed | Type: Observational
Sponsor: Pfizer's Upjohn has merged with Mylan to form Viatris Inc. (Industry)
Responsible Party: Sponsor
Organization: Pfizer (Industry)
Other Study IDs: A2581178
Record Dates: First submitted 2009-01-23; First posted 2009-01-26 (Estimated); Results first posted 2012-03-22 (Estimated); Last update posted 2021-02-21 (Actual); Status verified 2021-02

CONDITIONS: Hyperlipidemia
MeSH Terms: conditions — Hyperlipidemias

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Hyperlipidemic Patients
  Interventions: Device: Lipid Self Test

INTERVENTIONS:
Device: Lipid Self Test — Self test for lipid levels, twice during study period

SUMMARY:
It is a prospective observational study.

Patients will be high risk patients (for developing cardiovascular events) that are treated with a statin. Patients will be enrolled at a normal clinic visit and provided with a small box containing info about the disease, a LDL self-test and two questionnaires. They will test themselves for LDL at home between normal clinic visits (normally 12 months interval) and note their value. In the end of the study all patients will fill out a questionnaire with questions if the tests and info have raised their awareness of the disease as well if their motivation to be compliant has increased.

We want to look at the possibility to put more responsibility for treatment and for reaching treatment goals on the patients since there's a big problem with compliance in this group of patients.

DETAILED DESCRIPTION:
Consecutive patient sampling

ELIGIBILITY:
Inclusion Criteria:

* Aged 18 years or older and able to understand and sign the informed consent form.

  * Patients diagnosed with hyperlipidemia and a very high risk developing cardiovascular disease prescribed statin treatment according to clinical praxis and the recommendations set forth in the MPA national guideline for treatment of hyperlipidemia.

Exclusion Criteria:

* Patients contraindicated for statin treatment according to market authorization for these drugs should be excluded from the study.
* Patients participating in other clinical trials or non-interventional studies.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Aged 18 years or older and able to understand and sign the informed consent form.
  • Patients diagnosed with hyperlipidemia and a very high risk developing cardiovascular disease prescribed statin treatment according to clinical praxis and the recommendations set forth in the MPA national guideline for treatment of hyperlipidemia.
Sampling Method: Probability Sample
Enrollment: 259 (Actual)
Dates: Start 2009-02; Primary Completion 2011-03 (Actual); Study Completion 2011-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (15):
- Sweden (15):
  - Pfizer Investigational Site, Åkersberga
  - Pfizer Investigational Site, Forshaga
  - Pfizer Investigational Site, Gothenburg
  - Pfizer Investigational Site, Höganäs
  - Pfizer Investigational Site, Jönköping
  - Pfizer Investigational Site, Lessebo
  - Pfizer Investigational Site, Lilla Edet
  - Pfizer Investigational Site, Limhamn
  - Pfizer Investigational Site, Malmo
  - Pfizer Investigational Site, Oviken
  - Pfizer Investigational Site, Partille
  - Pfizer Investigational Site, Stockholm
  - Pfizer Investigational Site, Täby
  - Pfizer Investigational Site, Trollhättan
  - Pfizer Investigational Site, Västerås

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A2581178&StudyName=Compliance%20With%20Treatment%20For%20Patients%20With%20Hyperlipidemia

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: A total of 259 participants were enrolled in the study, out of which 2 participants were not evaluated due to screening failure.
Groups:
- Statins: Participants with hyperlipidemia; high risk of developing cardiovascular disease and taking lipid lowering treatment (statins) were observed for 12 months.
Period: Overall Study
Arm/Group | Statins
Started | 257
Completed | 216
Not Completed | 41
Not completed — Death | 4
Not completed — Participant was missing | 1
Not completed — Other | 36

BASELINE CHARACTERISTICS:
Arm/Group | Statins
Number analyzed (Participants) | 257
Age, Continuous [Mean (Standard Deviation); unit: Years] | 65.4 (9.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 108
  Male | 149
Positive response on self -estimated treatment compliance [Number; unit: Percentage of participants] — Participants with "Yes" response to a question which stated "Have you been taking at least 90 percentage (%) of your medication for hyperlipidemia?"
  Percentage of participants | 94.2
Low-density lipoprotein (LDL) lower than 2.5 millimole/liter (mmol/L) [Number; unit: Percentage of participants] — LDL levels were self-assessed by participants using CARE diagnostica LDL-cholesterol test. The targeted level of LDL was lower than 2.5 mmol/L.
  Percentage of participants | 30.7

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Positive Response on Increased Motivation Using a Self-test at Month 12
Description: Participants with "Yes" response to a question which stated "The self-test have increased my motivation for taking my medication for hyperlipidemia?". The self test done for assessment of LDL levels using CARE diagnostica LDL-cholesterol test.
Time Frame: Month 12
Population: The Full Analysis Set (FAS) included all enrolled participants who met all inclusion criteria.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Statins
Number analyzed (Participants) | 257
Percentage of participants | 36.2 [30.3 to 42.4]

2. Primary Outcome: Percentage of Participants With Positive Response on Increased Motivation After Awareness at Month 12
Description: Participants with "Yes" response to a question which stated "The awareness of my disease has increased my motivation for taking my medication for hyperlipidemia?".
Time Frame: Month 12
Population: The FAS included all enrolled participants who met all inclusion criteria.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Statins
Number analyzed (Participants) | 257
Percentage of participants | 54.9 [48.6 to 61.1]

3. Primary Outcome: Percentage of Participants With Positive Response on Self-estimated Treatment Compliance at Week 8
Description: Participants with "Yes" response to a question which stated "Have you been taking at least 90% of your medication for hyperlipidemia?".
Time Frame: Week 8
Population: The FAS included all enrolled participants who met all inclusion criteria.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Statins
Number analyzed (Participants) | 257
Percentage of participants | 74.3 [68.5 to 79.6]

4. Primary Outcome: Percentage of Participants With Positive Response on Self-estimated Treatment Compliance at Month 6
Description: as for outcome 3
Time Frame: Month 6
Population: The FAS included all enrolled participants who met all inclusion criteria.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Statins
Number analyzed (Participants) | 257
Percentage of participants | 61.1 [54.8 to 67.1]

5. Primary Outcome: Percentage of Participants With Positive Response on Self-estimated Treatment Compliance at Month 12
Description: as for outcome 3
Time Frame: Month 12
Population: The FAS included all enrolled participants who met all inclusion criteria.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Statins
Number analyzed (Participants) | 257
Percentage of participants | 75.9 [70.2 to 81.0]

6. Primary Outcome: Percentage of Participants With LDL Lower Than 2.5 mmol/L at Week 8
Description: LDL levels were self-assessed by participants using CARE diagnostica LDL-cholesterol test.
Time Frame: Week 8
Population: The FAS included all enrolled participants who met all inclusion criteria.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Statins
Number analyzed (Participants) | 257
Percentage of participants | 9.3 [6.1 to 13.6]

7. Primary Outcome: Percentage of Participants With LDL Lower Than 2.5 mmol/L at Month 6
Description: LDL levels were self-assessed by participants using CARE diagnostica LDL-cholesterol test.
Time Frame: Month 6
Population: The FAS included all enrolled participants who met all inclusion criteria.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Statins
Number analyzed (Participants) | 257
Percentage of participants | 8.2 [5.1 to 12.2]

8. Primary Outcome: Percentage of Participants With LDL Lower Than 2.5 mmol/L at Month 12
Description: LDL levels were self-assessed by participants using CARE diagnostica LDL-cholesterol test.
Time Frame: Month 12
Population: The FAS included all enrolled participants who met all inclusion criteria.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Statins
Number analyzed (Participants) | 257
Percentage of participants | 51.4 [47.8 to 60.3]

9. Primary Outcome: Percentage of Participants With Response Achieving Targeted LDL-cholesterol Level at Week 8
Description: Participants with "Yes" or "No" responses to a question which stated "Have you reached your target LDL-cholesterol level?". LDL levels were self-assessed by participants using CARE diagnostica LDL-cholesterol test.
Time Frame: Week 8
Population: The FAS included all enrolled participants who met all inclusion criteria.
Measure: Number; unit: Percentage of participants
Arm/Group | Statins
Number analyzed (Participants) | 257
Percentage of participants
  Yes | 14.8
  No | 18.3

10. Primary Outcome: Percentage of Participants With Response Achieving Targeted LDL-cholesterol Level at Month 6
Description: as for outcome 9
Time Frame: Month 6
Population: The FAS included all enrolled participants who met all inclusion criteria.
Measure: Number; unit: Percentage of participants
Arm/Group | Statins
Number analyzed (Participants) | 257
Percentage of participants
  Yes | 14.0
  No | 10.1

11. Primary Outcome: Percentage of Participants With Response Achieving Targeted LDL-cholesterol Level at Month 12
Description: as for outcome 9
Time Frame: Month 12
Population: The FAS included all enrolled participants who met all inclusion criteria.
Measure: Number; unit: Percentage of participants
Arm/Group | Statins
Number analyzed (Participants) | 257
Percentage of participants
  Yes | 31.9
  No | 13.6

ADVERSE EVENTS:
Description: The same event may appear as both an AE and a SAE. However, what is presented are distinct events. An event may be categorized as serious in one subject and as nonserious in another subject, or one subject may have experienced both a serious and nonserious event during the study.
Arm/Group | Statins
Serious Adverse Events (participants affected / at risk) | 7/259
Other Adverse Events (participants affected / at risk) | 0/259
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Statins (N=259)
Acute myocardial infarction (Cardiac disorders) | 1
Angina pectoris (Cardiac disorders) | 1
Worsening of angina pectoris (Cardiac disorders) | 1
Chest pain (General disorders) | 1
Death (General disorders) | 1
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Pancreatic cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Rectal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.